CLINICAL TRIAL: NCT00001998
Title: Pharmacokinetics of Nystatin LF I.V. in Patients With Acquired Immune Deficiency Syndrome-Related Complex (ARC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Argus Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 103A; AR-90-01-002
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-11

CONDITIONS: HIV Infections
Keywords: Nystatin; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Nystatin

INTERVENTIONS:
Drug: Nystatin

SUMMARY:
To define the pharmacokinetic characteristics of Nystatin LF IV (intravenous) in human subjects with AIDS-related complex (ARC) after administration of a single IV dose at each of 4 dose levels.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* Positive HIV antibody test.
* Diagnosis of AIDS-related complex (ARC).
* CD4+ cell count between 100 and 300 cells/mm3.
* Estimated life expectancy of at least 6 months.
* Normal neurological status.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Active opportunistic infection requiring ongoing therapy except patients being treated topically for oral thrush.

Patients with the following are excluded:

* Active opportunistic infection.
* Known hypersensitivity to polyene antibiotics.
* Unwillingness to sign an informed consent or to be in compliance of protocol requirements.

Prior Medication:

Excluded within 72 hours of study entry:

* Biologic response modifier agents.
* Corticosteroids.
* Cytotoxic chemotherapeutic agents.
* Potential nephrotoxins.
* Potential neutropenic agents.
* Rifampin or rifampin derivatives.
* Systemic anti-infectives.
* Phenytoin or barbiturates (inducers of microsomal enzymes).
* All systemic medications.

Prior Treatment:

Excluded within 72 hours prior to study entry:

* Radiation therapy.

Active alcohol or drug abuse unless they have been off drugs and/or alcohol for two weeks prior to start of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Twelve Oaks Hosp, Houston, Texas, United States

REFERENCES:
- [Background] Rios A, Crofoot GE, Lenk R, Hayman A, Rosenblum M, Lopez-Berestein G. A phase 1 single dose safety evaluation and pharmacokinetic (Pkc) study of nystatin-liposomal formulation nystatin-LF i.v. in patients with HIV infection. Int Conf AIDS. 1992 Jul 19-24;8(3):127 (abstract no PuB 7473)